CLINICAL TRIAL: NCT05227027
Title: Influence of a Game Embedded in a Smartphone App for Smoking Cessation on User Engagement: A Randomized Pilot Trial
Brief Title: Pilot Trial of a Game Embedded in a Smartphone App for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute on Aging (NIA) (NIH); University of California, Berkeley (Other); Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 19-29335; NCI-2021-07004 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30AG012839 (NIH); R21CA238301 (NIH)
Record Dates: First submitted 2022-01-26; First posted 2022-02-07 (Actual); Results first posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-11

CONDITIONS: Cigarette Smoking-Related Carcinoma
MeSH Terms: interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Education plus game module (Experimental): Participants receive an educational intervention through the Smoke Free application with the embedded game module. Participants complete questionnaires and may undergo saliva sample collection, if they report being smoke-free on follow-up.
  Interventions: Behavioral: Game Module; Behavioral: Smoke Free smartphone application
- Education module only (Active Comparator): Participants receive an educational intervention through the Smoke Free application only (core app only). Participants complete questionnaires and may undergo saliva sample collection, if they report being smoke-free on follow-up.
  Interventions: Behavioral: Smoke Free smartphone application

INTERVENTIONS:
Behavioral: Game Module — Receive access to the the game module through the free, 'Smoke Free' smartphone application
  Other Names: In-application game module
  Arms: Education plus game module
Behavioral: Smoke Free smartphone application — Receive educational intervention through the free 'Smoke Free' smartphone application (core version of the app)
  Other Names: Educational intervention

SUMMARY:
This study evaluates the effects of a video game embedded in a commercially available mobile application (app) for smoking cessation. Smokers are increasingly turning to mobile health apps for assistance with quitting smoking, and there is a critical need for strategies to engage app users to increase retention and efficacy. Video games are designed to increase users' motivation and engagement, which in turn may increase their exposure and adherence to a smoking cessation program. The hypothesis is that the game increases engagement, retention, and smoking abstinence rates compared with a core version of the app without the game. A two-arm individually randomized pilot trial of 500 adult smokers will test this hypothesis, comparing outcomes for participants randomized to receive the core app plus embedded game with participants randomized to receive the core app only. Primary outcomes relate to user engagement with the app. Secondary outcomes relate to user engagement, efficacy (smoking abstinence), and user satisfaction.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Augment an existing smartphone cessation app for smoking cessation with a video game to increase user engagement.

II. Test the feasibility, engagement, and early efficacy of the 'gamified' app, compared to one without gamification.

OUTLINE:

Participants are recruited through the Smoke Free smartphone app and randomized to 1 of 2 arms.

ARM I: Participants receive an educational intervention through the Smoke Free application (core app) with the embedded video game module. Participants complete questionnaires and may undergo saliva sample collection, if they report being smoke-free on follow-up.

ARM II: Participants receive an educational intervention through the Smoke Free application without the video game module (core app only). Participants complete questionnaires and may undergo saliva sample collection, if they report being smoke-free on follow-up.

ELIGIBILITY:
Inclusion criteria:

1. Provides electronic informed consent.
2. Male or female, aged 18 and older
3. Has downloaded and opened the Smoke Free app
4. A smoker of at least 1 cigarette per day
5. Plans to quit smoking within the next 7 days
6. Speaks, reads, and writes English
7. Lives in the United States

Exclusion criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin White, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] White JS, Salem MK, Toussaert S, Westmaas JL, Raiff BR, Crane D, Warrender E, Lyles C, Abroms L, Thrul J. Developing a Game (Inner Dragon) Within a Leading Smartphone App for Smoking Cessation: Design and Feasibility Evaluation Study. JMIR Serious Games. 2023 Aug 11;11:e46602. doi: 10.2196/46602. PMID 37566442
- [Derived] White JS, Toussaert S, Raiff BR, Salem MK, Chiang AY, Crane D, Warrender E, Lyles CR, Abroms LC, Westmaas JL, Thrul J. Evaluating the Impact of a Game (Inner Dragon) on User Engagement Within a Leading Smartphone App for Smoking Cessation: Randomized Controlled Trial. J Med Internet Res. 2024 Oct 30;26:e57839. doi: 10.2196/57839. PMID 39475840

RESULTS

PARTICIPANT FLOW:
Groups:
- Educational Intervention Plus Game Module: Participants receive free access to an educational intervention consisting of the core features of the Smoke Free application, as well as the integrated game module. Participants complete questionnaires and are invited to completed remote saliva sample collection if they report being smoke-free at follow-up.
  Smoke Free educational intervention: Receive free access to core features of the Smoke Free smartphone application, including a calculator that tracks time elapsed since quitting smoking, progress indicators regarding predicted health improvements, daily tasks to avoid and resist urges to smoke, and a text-based chatbot that delivers smoking cessation guidance.
  Game module: Receive free access to the the Inner Dragon game module integrated into the Smoke Free smartphone application. In the Inner Dragon game, users care for a customizable pet dragon. that "evolves" in tandem with the user's progress in quitting smoking. The game includes several key features: 1) the dragon hatches on the user's quit day and evolves every 7 days to unlock new attributes and powers; 2) users earn experience points by using selected core app features; 3) users maintain "care meters" that change when the dragon is fed or pet; 4) the game provides tools for the user to better cope with the challenges of withdrawal, such as a breathing exercise to provide calmness and a memory minigame as a distraction; and 5) users can asynchronously interact with other users' dragons in a "dragon park."
- Educational Intervention Only: Participants receive free access to an educational intervention consisting of the core features of the Smoke Free application only. Participants complete questionnaires and are invited to completed remote saliva sample collection if they report being smoke-free at follow-up.
  Smoke Free educational intervention: Receive free access to core features of the Smoke Free smartphone application, including a calculator that tracks time elapsed since quitting smoking, progress indicators regarding predicted health improvements, daily tasks to avoid and resist urges to smoke, and a text-based chatbot that delivers smoking cessation guidance.
Period: Overall Study
Arm/Group | Educational Intervention Plus Game Module | Educational Intervention Only
Started | 251 | 249
Completed | 241 | 238
Not Completed | 10 | 11
Not completed — Did not finish the onboarding process within the Smoke Free app prior to learning their allocation | 10 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Educational Intervention Plus Game Module | Educational Intervention Only | Total
Number analyzed (Participants) | 241 | 238 | 479
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38 [29 to 47] | 35 [28 to 47] | 36 [29 to 47]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 177 | 181 | 358
  Gender: Male | 59 | 55 | 114
  Gender: Non-binary or other | 5 | 2 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race and ethnicity: Non-Hispanic White | 186 | 182 | 368
  Race and ethnicity: Non-Hispanic Black | 22 | 26 | 48
  Race and ethnicity: Hispanic | 19 | 9 | 28
  Race and ethnicity: Other | 14 | 21 | 35
Educational attainment [Count of Participants; unit: Participants]
  High school diploma or less | 45 | 55 | 100
  Some college or technical school | 93 | 84 | 177
  Bachelor's or associate degree | 83 | 68 | 151
  Graduate degree | 20 | 31 | 51
Household income, categorical [Count of Participants; unit: Participants]
  Less than $20,000 | 35 | 35 | 70
  Between $20,000 and $40,000 | 63 | 65 | 128
  Between $40,000 and $60,000 | 51 | 51 | 102
  Between $60,000 and $80,000 | 32 | 24 | 56
  Between $80,000 and $100,000 | 21 | 18 | 39
  More than $100,000 | 39 | 45 | 84
Cigarettes per day [Median (Inter-Quartile Range); unit: cigarettes] | 15 [10 to 20] | 15 [10 to 20] | 15 [10 to 20]
Fagerström Test for Nicotine Dependence [Median (Inter-Quartile Range); unit: units on a scale] — Fagerström Test for Nicotine Dependence is a 6-item measure of nicotine dependence. It has a scale range from 0 (low dependence) to 10 (high dependence). The total score is reported.
  units on a scale | 5 [4 to 7] | 5 [3 to 7] | 5 [4 to 7]
Past quit attempts [Median (Inter-Quartile Range); unit: attempts] | 4 [2 to 9] | 4 [2 to 8] | 4 [2 to 9]
Years since initiated smoking [Median (Inter-Quartile Range); unit: years] | 19 [11 to 29] | 16 [10 to 28] | 18 [10 to 29]
Used electronic nicotine device systems in last 30 days [Count of Participants; unit: Participants] | 57 | 61 | 118
Used nicotine replacmeent therapy in last 30 days [Count of Participants; unit: Participants] | 56 | 43 | 99
Frequency played video games in last 6 months [Count of Participants; unit: Participants]
  Not at all | 57 | 59 | 116
  Less than once a month | 36 | 25 | 61
  At least monthly but not weekly | 26 | 25 | 51
  At least weekly but not every day | 49 | 40 | 89
  Every day | 73 | 89 | 162

OUTCOME MEASURES:

1. Primary Outcome: Number of Unique App Sessions
Description: Number of times the app was opened; passively collected by the app and averaged in analysis to calculate mean number of app opens by study group over the study period. A new session is defined as use of the app after at least 30 minutes of inactivity.
Time Frame: Enrollment through 56 days after participant's selected quit date (56 to 63 days total)
Measure: Mean (Standard Deviation); unit: number of sessions
Arm/Group | Educational Intervention Plus Game Module | Educational Intervention Only
Number analyzed (Participants) | 241 | 238
number of sessions | 29.6 (36.5) | 24.3 (37.9)

2. Primary Outcome: Minutes of App Usage Per Session
Description: Passively collected by the app and averaged in analysis among those with a session to calculate mean number of minutes of usage per session by study group.
Time Frame: Enrollment through 56 days after participant's selected quit date (56 to 63 days total)
Measure: Mean (Standard Deviation); unit: minutes per session
Arm/Group | Educational Intervention Plus Game Module | Educational Intervention Only
Number analyzed (Participants) | 241 | 238
minutes per session | 6.9 (5.4) | 6.1 (5.2)

3. Secondary Outcome: Unique Days With at Least One App Session
Description: Number of unique days with at least one app session, passively collected by the app and averaged by study group.
Time Frame: Enrollment through 56 days after participant's selected quit date (56 to 63 days total)
Measure: Mean (Standard Deviation); unit: days with a session
Arm/Group | Educational Intervention Plus Game Module | Educational Intervention Only
Number analyzed (Participants) | 241 | 238
days with a session | 14.3 (15.3) | 11.9 (13.3)

4. Secondary Outcome: Self-reported 7-day Point-prevalence Abstinence at 2 Months
Description: Proportion of participants who self-report having abstained for the prior 7 days during the 2-month follow-up assessment, assuming missing = smoking.
Time Frame: 56 days after participant's selected quit date (56 to 63 days after enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Educational Intervention Plus Game Module | Educational Intervention Only
Number analyzed (Participants) | 241 | 238
Participants | 94 | 101

5. Secondary Outcome: Self-reported 30-day Point-prevalence Abstinence at 2 Months
Description: Proportion of participants who who self-report having abstained for the prior 30 days during the 2-month follow-up assessment, assuming missing = smoking.
Time Frame: 56 days after participant's selected quit date (56 to 63 days after enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Educational Intervention Plus Game Module | Educational Intervention Only
Number analyzed (Participants) | 241 | 238
Participants | 54 | 50

6. Secondary Outcome: Satisfaction With App
Description: Rating of satisfaction with assigned app on a 5-point Likert scale from "Not at all" (1) to "Extremely" (5), assessed in the 2-month follow-up questionnaire. The measure is averaged by study group.
Time Frame: 56 days after participant's selected quit date (56 to 63 days after enrollment)
Population: Only those participants who completed the follow-up questionnaire are included in the analysis population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Intervention Plus Game Module | Educational Intervention Only
Number analyzed (Participants) | 144 | 127
units on a scale | 3.7 (1.0) | 3.7 (1.1)

7. Secondary Outcome: Satisfaction With Game (Intervention Group Only)
Description: Rating of satisfaction with the game on a 5-point Likert scale from "Not at all" (1) to "Extremely" (5), assessed in the 2-month follow-up questionnaire. The measure is averaged for the intervention group.
Time Frame: 56 days after participant's selected quit date (56 to 63 days after enrollment)
Population: Only those participants in the intervention group who completed the follow-up questionnaire are included in the analysis population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Intervention Plus Game Module | Educational Intervention Only
Number analyzed (Participants) | 84 | 0
units on a scale | 3.3 (1.4) |

8. Other Pre Specified Outcome: Biochemically Verified 7-day Point-prevalence Abstinence at 2 Months
Description: Proportion of participants who who self-report having abstained for the prior 7 days during the 2-month follow-up assessment, verified by saliva cotinine test, assuming missing = smoking. Averaged by study group. Recoded to 0 if the person reported having smoked during the same 7-day window during repeated measurement of daily smoking in the app.
Time Frame: 56 days after participant's selected quit date (56 to 63 days after enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Educational Intervention Plus Game Module | Educational Intervention Only
Number analyzed (Participants) | 241 | 238
Participants | 27 | 37

9. Other Pre Specified Outcome: Biochemically Verified 30-day Point-prevalence Abstinence at 2 Months
Description: Proportion of participants who who self-report having abstained for the prior 30 days during the 2-month follow-up assessment, verified by saliva cotinine test, assuming missing = smoking. Averaged by study group. Recoded to 0 if the person reported having smoked during the same 30-day window during repeated measurement of daily smoking in the app.
Time Frame: 56 days after participant's selected quit date (56 to 63 days after enrollment)
Measure: Count of Participants; unit: Participants
Arm/Group | Educational Intervention Plus Game Module | Educational Intervention Only
Number analyzed (Participants) | 241 | 238
Participants | 19 | 31

10. Other Pre Specified Outcome: Repeated 1-day Point-prevalence Smoking Abstinence
Description: Proportion of days in which participants self-report having abstained in the last 24 hours, collected via a pop-up box that appears the first time each day a participant opens the app. Averaged by study group.
Time Frame: During the 56 days after participant's selected quit date
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Educational Intervention Plus Game Module | Educational Intervention Only
Number analyzed (Participants) | 241 | 238
percentage of days | 17.3 (25.6) | 12.4 (21.3)

11. Other Pre Specified Outcome: Program Adherence (Index of Core Feature Use)
Description: Number of non-game (core app) activities completed in the app by activity type: passively collected by the app to assess number of times the participant completed the following activity types: reported a craving, recorded a diary, completed a mission, read a tip, used the chatbot.
Time Frame: Enrollment through 56 days after participant's selected quit date (56 to 63 days total)
Measure: Mean (Standard Deviation); unit: number of core features used
Arm/Group | Educational Intervention Plus Game Module | Educational Intervention Only
Number analyzed (Participants) | 241 | 238
number of core features used | 19.0 (28.2) | 15.6 (29.1)

12. Other Pre Specified Outcome: Gifts Unlocked (Intervention Group Only)
Description: Number of in-game gifts unlocked during the study period (intervention group only); a summary measure of intensity of engagement (dose of treatment) of the app; passively collected by the app.
Time Frame: Enrollment through 56 days after participant's selected quit date (56 to 63 days total)
Population: In-game gifts available for intervention group only.
Measure: Mean (Standard Deviation); unit: number of gifts unlocked
Arm/Group | Educational Intervention Plus Game Module | Educational Intervention Only
Number analyzed (Participants) | 241 | 0
number of gifts unlocked | 3.3 (6.9) |

13. Other Pre Specified Outcome: Game Activities (Intervention Group Only)
Description: Number of game activities completed in the app by activity type; passively collected by the app to assess number of times the participant completed the following activity types: navigated to the game dashboard, completed each pet care activity (breathing exercise, feeding, washing, memory mini-game), visited the park, entered the dragon guide.
Time Frame: Enrollment through 56 days after participant's selected quit date (56 to 63 days total)
Population: Applicable to intervention group only.
Measure: Mean (Standard Deviation); unit: number of game features used
Arm/Group | Educational Intervention Plus Game Module | Educational Intervention Only
Number analyzed (Participants) | 241 | 0
number of game features used | 123.1 (285.0) |

14. Other Pre Specified Outcome: Recommends App to Friend
Description: Rating of whether would recommend assigned app to a friend on a 5-point Likert scale from "Not at all" (1) to "Extremely" (5), assessed in the 2-month follow-up questionnaire. The measure is averaged by study group.
Time Frame: 56 days after participant's selected quit date (56 to 63 days after enrollment)
Population: Only those participants who completed the follow-up questionnaire are included in the analysis population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Intervention Plus Game Module | Educational Intervention Only
Number analyzed (Participants) | 144 | 127
units on a scale | 3.8 (1.1) | 4.0 (1.1)

15. Other Pre Specified Outcome: Motivation to Quit
Description: Motivation to quit, reported on a 10-point scale from not at all motivated (0) to very unmotivated (10) and assessed in the 2-month follow-up.
Time Frame: 56 days after participant's selected quit date (56 to 63 days after enrollment)
Population: Only those participants who completed the question in the follow-up questionnaire are included in the analysis population. A programming error led to missing data for most respondents who reported having continued to smoke.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Intervention Plus Game Module | Educational Intervention Only
Number analyzed (Participants) | 73 | 71
units on a scale | 9.3 (1.3) | 9.4 (1.5)

16. Other Pre Specified Outcome: Digital Therapeutic Alliance
Description: The measure includes items from the Bonding and Confidence subscales from the Mobile Agnew Relationship Measure, a scale of digital therapeutic alliance. Two items from each of the Bonding and Confidence subscales were included. Each item was asked on a 4-point Likert scale from strongly disagree (1) to strongly agree (4). The subscale items were combined to give a total possible score of 16 and a range of 4 (low alliance) to 16 (high alliance). The measure is averaged by study group. Assessed in the 2-month follow-up.
Time Frame: 56 days after participant's selected quit date (56 to 63 days after enrollment)
Population: Only those participants who completed the questions in the follow-up questionnaire are included in the analysis population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Intervention Plus Game Module | Educational Intervention Only
Number analyzed (Participants) | 150 | 129
units on a scale | 12.7 (2.2) | 12.8 (2.5)

ADVERSE EVENTS:
Time Frame: 63 days after enrollment
Description: Adverse events were reported based on survey responses to "Did you experience any negative, unpleasant, unwanted, or otherwise unexpected side effects as a result of participating in this trial?"
Arm/Group | Educational Intervention Plus Game Module | Educational Intervention Only
All-Cause Mortality (participants affected / at risk) | 0/241 | 0/238
Serious Adverse Events (participants affected / at risk) | 0/241 | 0/238
Other Adverse Events (participants affected / at risk) | 3/241 | 7/239
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Educational Intervention Plus Game Module (N=241) | Educational Intervention Only (N=239)
Anxious or depressed (Psychiatric disorders) | 1 | 3 — Reported being anxious or depressed
Feelings of withdrawal, craving, or irritability (Psychiatric disorders) | 1 | 4 — Reported feelings of withdrawal, craving, or irritability
Constipation (Gastrointestinal disorders) | 1 | 0 — Reported constipation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/27/NCT05227027/Prot_SAP_001.pdf
  • Informed Consent Form (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT05227027/ICF_000.pdf